CLINICAL TRIAL: NCT02766439
Title: the First People's Hospital of Chenzhou
Brief Title: Rhupus Syndrome and Efficacy of Etanercept Treatment
Status: Completed | Type: Observational
Sponsor: Yang Beibei (Other)
Responsible Party: Sponsor-Investigator, Yang Beibei, the First People's Hospital of Chenzhou, First People's Hospital of Chenzhou
Organization: First People's Hospital of Chenzhou (Other)
Other Study IDs: 201233-004
Record Dates: First submitted 2016-05-06; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Rhupus Syndrome, Etanercept
MeSH Terms: conditions — rhupus syndrome | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rhupus syndrome, SLE without RA: Rhupus syndrome, SLE without RA
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — 25-mg etanercept injection subcutaneously twice a week
  Other Names: TNFа blockade

SUMMARY:
between March 2013 and March 2014, Rhupus patients were enrolled to receive a 25-mg etanercept injection subcutaneously twice a week. The follow-up time of the study was 24 weeks.

DETAILED DESCRIPTION:
between March 2013 and March 2014, patients who were unresponsive to therapy with corticosteroid and disease-modifying antirheumatic drugs (DMARDs), with a Disease Activity Score in 28 Joints (DAS28) >5.1 were enrolled to receive a 25-mg etanercept injection subcutaneously twice a week. The follow-up time of the study was 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Rhupus patients who were unresponsive to therapy with corticosteroid and disease-modifying antirheumatic drugs (DMARDs), with a Disease Activity Score in 28 Joints (DAS28) >5.1

Exclusion Criteria:

- those who had participated in other studies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were unresponsive to therapy with corticosteroid and disease-modifying antirheumatic drugs (DMARDs), with a Disease Activity Score in 28 Joints (DAS28) >5.1 were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score in 28 Joints (DAS28) | 24 week

IPD SHARING:
Plan to Share IPD: Undecided